CLINICAL TRIAL: NCT07259824
Title: Evaluation of the Effectiveness of Serratus Posterior Superior Intercostal Plane Block in Perioperative Pain Management in Patients Undergoing Minimally Invasive Cardiac Surgery
Brief Title: SPSIP Block and Opioid Use After MICS
Acronym: SPSIPB-MICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nisan Özsan, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NisanOzsan
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Valvular Disease; Minimally Invasive Cardiac Surgery; Postoperative Pain Management; Serratus Posterior Superior Intercostal Plane Block
Keywords: postoperative pain management; minimally invasive cardiac surgery; serratus posterior superior intercostal plane block; opioid consumption
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, parallel-group clinical trial conducted at a single center. Eligible patients scheduled for minimally invasive cardiac surgery will be randomly assigned in a 1:1 ratio to receive either the Serratus Posterior Superior Intercostal Plane Block (SPSIPB) in addition to standard analgesia or standard analgesia alone. Both groups will be managed and evaluated under the same perioperative protocol, and outcomes will be assessed by blinded observers.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The anesthesiologist performing the block will be aware of group allocation, while the patients and the anesthesiologist responsible for postoperative data collection will remain blinded to the intervention. Pain assessments and other outcome measurements will be conducted by a blinded senior anesthesia resident who is unaware of which treatment each patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIPB Group (Experimental): Patients in this group will receive ultrasound-guided Serratus Posterior Superior Intercostal Plane Block (SPSIPB) with 30 mL of 0.25% bupivacaine in addition to standard anesthesia and analgesia.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block (SPSIPB)
- Sham Block Group (Sham Comparator): Patients in this group will undergo the same ultrasound-guided block procedure using identical technique and needle placement, but 30 mL of normal saline will be injected instead of local anesthetic. All other anesthesia and analgesia protocols will be identical to the experimental group.
  Interventions: Procedure: Sham Serratus Posterior Superior Intercostal Plane Block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block (SPSIPB) — The SPSIPB will be performed under ultrasound guidance using an in-plane technique. The needle will be advanced into the fascial plane between the serratus posterior superior and intercostal muscles at the 2nd-3rd intercostal level, and 30 mL of 0.25% bupivacaine will be injected unilaterally on the surgical side. This procedure will be applied in addition to standard anesthesia and analgesia.
  Arms: SPSIPB Group
Procedure: Sham Serratus Posterior Superior Intercostal Plane Block — The same ultrasound-guided procedure will be performed using identical technique and needle placement, but 30 mL of normal saline will be injected instead of local anesthetic. This sham block will be performed to maintain blinding, while all other anesthesia and analgesia protocols will be identical to the experimental group.
  Arms: Sham Block Group

SUMMARY:
This prospective, randomized, controlled, single-center clinical study aims to evaluate the effectiveness of the Serratus Posterior Superior Intercostal Plane Block (SPSIPB) in perioperative pain management among patients undergoing minimally invasive cardiac surgery (MICS). A total of 50 patients undergoing MICS will be randomized into two groups: one receiving standard analgesia plus ultrasound-guided SPSIPB with 30 mL of 0.25% bupivacaine, and a control group receiving standard analgesia only. The primary outcome is total postoperative opioid consumption within 24 hours. Secondary outcomes include postoperative pain scores, extubation time, block-related complications, and recovery parameters such as early mobilization, oral intake, Modified radiological atelectasis score and Quality of Recovery-15 scores.

DETAILED DESCRIPTION:
Minimally invasive cardiac surgery (MICS) is increasingly performed as an alternative to traditional sternotomy-based procedures, providing benefits such as shorter recovery time, reduced hospital stay, and improved cosmetic outcomes. However, despite smaller incisions, patients frequently experience moderate to severe postoperative pain due to rib, pleural, and intercostal nerve injury. Uncontrolled pain may impair respiratory function, delay mobilization, and increase postoperative complications, including chronic post-thoracotomy pain.

Regional anesthesia techniques play an important role in multimodal analgesia after MICS, but the optimal approach remains uncertain. Thoracic epidural and paravertebral blocks have been widely used but are often limited by safety concerns in anticoagulated patients. Recently, ultrasound-guided interfascial plane blocks have gained attention due to their simplicity and low complication rates. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB), first described in 2023, targets the fascial plane between the serratus posterior superior and intercostal muscles, typically at the second or third intercostal level, and provides broad sensory coverage from C3 to T10 dermatomes. To date, there is no published study investigating its use for pain control in MICS.

This study will be conducted at Ankara Bilkent City Hospital as a prospective, randomized, controlled, single-center clinical trial. A total of 50 patients (25 per group) aged 18-75 years (ASA II-III) scheduled for MICS will be enrolled after obtaining informed consent. Participants will be randomly assigned (1:1) to one of two groups using a computer-based randomization method:

Group SPSIPB (n=25): Standard anesthesia and analgesia + ultrasound-guided SPSIPB with 30 mL of 0.25% bupivacaine (unilateral, on the surgical side).

Group Control (n=25): Standard anesthesia and analgesia only. All patients will receive intravenous tramadol (1 mg/kg) and paracetamol (1 g) at the end of surgery. Postoperative patient-controlled analgesia (PCA) with tramadol (15 mg bolus, 15-min lockout, no basal infusion) will be used in both groups. Rescue morphine (0.05 mg/kg) will be administered when NRS >4. Pain scores (NRS 0-10) will be recorded at 6, 12, and 24 hours postoperatively, both at rest and during deep breathing/coughing.

The primary outcome is total postoperative opioid consumption (morphine equivalent, mg) in the first 24 hours.

Secondary outcomes include intraoperative opioid use, postoperative pain scores, extubation time, block-related complications (e.g., pneumothorax, vascular puncture, hematoma, local anesthetic toxicity), postoperative recovery indicators (first oral intake, mobilization, respiratory function), Modified radiological atelectasis score, Quality of Recovery-15 (QoR-15) scores, and patient satisfaction.

All postoperative assessments will be performed by a blinded senior anesthesia resident unaware of group allocation. Statistical analysis will be conducted using SPSS v26. Continuous variables will be analyzed with the independent t-test or Mann-Whitney U test as appropriate; categorical variables will be evaluated with chi-square or Fisher's exact test. Repeated pain scores will be compared using repeated-measures ANOVA or Friedman test. A p value <0.05 will be considered statistically significant.

The study is expected to start in January 2026. The results may provide new evidence on the effectiveness and safety of SPSIPB for postoperative analgesia in minimally invasive cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for minimally invasive cardiac surgery (MICS)
* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) physical status II-III
* Body mass index (BMI) between 18 and 35 kg/m²
* Patients who provide written informed consent for participation

Exclusion Criteria:

* Known allergy or hypersensitivity to local anesthetics
* Coagulopathy or current anticoagulant therapy
* Pregnancy or breastfeeding
* Impaired consciousness or inability to communicate
* Failed or technically inadequate block
* Refusal to undergo the block procedure
* Cognitive or mental disorders preventing valid pain assessment
* Opioid intolerance or contraindication to opioid use
* Development of intraoperative or postoperative complications requiring reoperation, prolonged mechanical ventilation, or intensive care
* Incomplete postoperative data or patient withdrawal from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption within 24 hours after surgery | 24 hours postoperatively
  The total amount of opioids (converted to intravenous morphine equivalent, mg) administered during the first 24 postoperative hours will be recorded from the patient-controlled analgesia (PCA) device and rescue analgesic doses.

SECONDARY OUTCOMES:
Postoperative pain scores (NRS) | 6, 12, and 24 hours postoperatively
  Pain intensity will be assessed using the Numeric Rating Scale (0 = no pain, 10 = worst imaginable pain) at rest and during deep breathing/coughing.
Extubation time | Immediate postoperative period
  Time from the end of surgery to tracheal extubation (minutes).
Intraoperative opioid consumption | During surgery
  Total intraoperative opioid dose (converted to morphine equivalent, mg).
Block-related complications | Within 24 hours postoperatively
  Incidence of pneumothorax, vascular puncture, hematoma, local anesthetic systemic toxicity, or injection site pain.
Postoperative recovery parameters | Within 48 hours postoperatively
  Time to first oral intake, time to first mobilization assesment
Quality of Recovery (QoR-15) score | 24 and 48 hours postoperatively
  Patient recovery quality will be assessed using the validated QoR-15 questionnaire.The QoR-15 is a patient-reported outcome measure consisting of 15 items scored from 0 to 10. The total score ranges from 0 (extremely poor recovery) to 150 (excellent recovery), with higher scores reflecting better postoperative quality of recovery.
Modified Radiological Atelectasis Score | 24 and 48 hours postoperatively
  modified radiological atelectasis score will be evaluated at 24 and 48 hours after surgery. Each lung lobe, including the lingula, is scored from 0 (normal) to 3 (total atelectasis), with higher total scores indicating more severe atelectasis.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha A Demir, M.D., Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology and Reanimation, Professor of Aneshesiology; Aslıhan Aykut, M.D., Study Director — Ankara Bilkent City Hospital, Department of Anesthesiology and Reanimation, Associate Professor of Anesthesiology; Nisan Özsan, M.D., Study Chair — Ankara Bilkent City Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a single-center academic study. Individual participant data will not be shared publicly. Aggregate results will be reported in publication.

REFERENCES:
- [Background] Turan EI, Isik S, Baydemir AE, Sahin AS. Serratus posterior superior intercostal plane block for postoperative analgesia in clavicle surgeries: new indications for a novel block. Minerva Anestesiol. 2024 Nov;90(11):1058-1060. doi: 10.23736/S0375-9393.24.18275-2. Epub 2024 Aug 5. No abstract available. PMID 39101308
- [Background] Avci O, Gundogdu O, Balci F, Tekcan MN, Ozbey M. Efficacy of serratus posterior superior intercostal plane block (SPSIPB) on post-operative pain and total analgesic consumption in patients undergoing video-assisted thoracoscopic surgery (VATS): A double-blinded randomised controlled trial. Indian J Anaesth. 2023 Dec;67(12):1116-1122. doi: 10.4103/ija.ija_589_23. Epub 2023 Dec 13. PMID 38343684
- [Background] Shimizu C, Wakimoto M, Kita T. Efficacy of epidural anesthesia in minimally invasive cardiac surgery. Saudi J Anaesth. 2024 Oct-Dec;18(4):528-533. doi: 10.4103/sja.sja_334_24. Epub 2024 Oct 2. PMID 39600439
- [Background] Dost B, Turunc E, Aydin ME, Kaya C, Aykut A, Demir ZA, Narayanan M, De Cassai A. Pain Management in Minimally Invasive Cardiac Surgery: A Review of Current Clinical Evidence. Pain Ther. 2025 Jun;14(3):913-930. doi: 10.1007/s40122-025-00739-1. Epub 2025 Apr 24. PMID 40272720
- [Background] Piekarski F, Rohner M, Monsefi N, Bakhtiary F, Velten M. Anesthesia for Minimal Invasive Cardiac Surgery: The Bonn Heart Center Protocol. J Clin Med. 2024 Jul 5;13(13):3939. doi: 10.3390/jcm13133939. PMID 38999504